CLINICAL TRIAL: NCT05042115
Title: Osteopathic Manipulative Treatment Associated With Education About Pain and Clinical Hypnosis and Their Repercussions on Pain and Disability in Chronic Low Back Pain - Randomized Clinical Trial
Brief Title: Effects of Osteopathic Manipulative Treatment Associated With Pain Education and Clinical Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Docusse de Osteopatia e Terapia Manual (Network)
Collaborators: Universidade Estadual do Norte do Paraná (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43063621.3.0000.8123
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Educational Status; Hypnosis; Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Education in Pain Neuroscience through Clinical Hypnosis associated with Osteopathic Manipulative Treatment
Who Masked: Outcomes Assessor
Masking Description: A simple randomized sequence will be created through the website www.randomization.com by a collaborator external to the researchers directly involved in the research. After the initial assessment, the researcher will access the randomization envelope and the participant will be allocated to 1 of the 2 treatment groups. The allocation will be hidden using opaque envelopes, sealed, and identified by number. The researcher/evaluator will be blinded to the allocation of intervention groups. Given the nature of the study, it is impossible to blind the researcher/therapist and volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education in pain neurosciences and clinical hypnosis (Experimental): Pain neuroscience education and clinical hypnosis
  Interventions: Other: Education in pain neurosciences and clinical hypnosis
- Education in pain neurosciences and clinical hypnosis plus Osteopathic manipulative treatment (Active Comparator): Pain neuroscience education and clinical hypnosis, associated with osteopathic manipulative treatment
  Interventions: Other: Education in pain neurosciences and clinical hypnosis plus osteopathic manipulative treatment

INTERVENTIONS:
Other: Education in pain neurosciences and clinical hypnosis — Will be performed education in pain neurosciences and clinical hypnosis, in 4 sessions during 4 weeks
  Arms: Education in pain neurosciences and clinical hypnosis
Other: Education in pain neurosciences and clinical hypnosis plus osteopathic manipulative treatment — Will be performed education in pain neurosciences and clinical hypnosis, and only for this group will be delivered osteopathic manipulative treatment, in 4 sessions during 4 weeks
  Arms: Education in pain neurosciences and clinical hypnosis plus Osteopathic manipulative treatment

SUMMARY:
INTRODUCTION: Chronic low back pain (CLBD) is one of the major public health problems in the world. Given the complexity of the situation, complementary and alternative practices such as pain neuroscience education (PNE), clinical hypnosis (HC) and osteopathic manipulative treatment (OMT) are options for we manage these patients. OBJECTIVE: The aim of this study will be to evaluate the effects of OMT associated with PNE through HC on pain and disability in patients with CLBP compared to PNE and HC. MATERIALS AND METHODS: The study design will be a randomized clinical trial and 40 adults diagnosed with chronic low back pain will be recruited. Subjects will be randomized in two groups: the first group (G1) will be submitted to the PNE based on information from the book "Explain Pain" with hypnotic suggestions. Group 2 (G2) will receive PNE following the book "Explain Pain" with hypnotic suggestions associated with OMT. Volunteers will be evaluated by a blind researcher the interventions performed in the allocation of groups. The evaluation moments will be pre-intervention and immediately after the end of the last intervention for G1 and G2. Volunteers continued to be evaluated 4 weeks after completion of the protocols. Pain will be evaluated as the main outcome, being evaluated by the numerical pain scale. Pain will also be assessed by the pressure threshold using a pressure algometer device (Fnd-50, PIAB 50-n, Italy) in the lumbar region. Still as the main outcome, disability will be assessed using the Oswestry Disability Questionnaire. As secondary outcomes, the patient's global impression of improvement, central sensitization, biopsychosocial factors will be evaluated. The patient's global impression of improvement will be assessed using the Percentage of Improvement Scale with a score of -5 to +5; the Central Sensitization will be assessed using the Central Sensitization Questionnaire and the biopsychosocial factors using the Start Beck Toll questionnaire. In addition, the behavior of the autonomic nervous system will be evaluated through the Heart Rate Variability (HRV), which will be analyzed through linear methods, in the domains of time and frequency, and by geometric indices. The researcher/evaluator will be blinded to the allocation of intervention groups. Given the nature of the study, it is impossible to blind the researcher/therapist and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific Low Back Pain for at least 3 months
* Score on the numerical pain scale of at least 3 points

Exclusion Criteria:

* Data from participants with less than 95% of sinus beats
* Participants that present increased symptoms in any stages of the study
* Patients who are undergoing concomitant physical therapy treatment, patients with contraindications to exercise, smokers/alcoholics, severe vertebral or neural pathologies, previous spine surgeries, cardiorespiratory disease, LBP as a secondary complaint, pregnancy, hearing problems, or illiteracy patients, not will are able to participate the protocol.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Pain perception | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  The Pain suffered in the last week will be assessed by the Numerical pain scale, with a range of 0 - 10
Pain pressure threshold | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  Pain will be assessed by the pressure threshold using a pressure algometer device in the lumbar region. The assessment will be conducted specifically in the paravertebral muscles bilaterally at levels L1 to L5.
Disability | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  Disability will be assessed using the Oswestry Disability Questionnaire

SECONDARY OUTCOMES:
Patient's global impression of improvement | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  The patient's global impression of improvement will be assessed using the Percentage of Improvement Scale with a score of -5 to +5
Central Sensitization and biopsychosocial factors | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  The Central Sensitization Questionnaire and the biopsychosocial factors will be assessed using the Start Beck Toll questionnaire
Heart Rate Variability | T0= before the protocol; T1= until 24 hours after the end protocol; T2= four weeks after end protocols
  Heart Rate Variability, which will be analyzed through linear methods, in the domains of time and frequency, and by geometric indices

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Kastelianne, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared by request
Supporting Information: Study Protocol, SAP
Time Frame: After one year from publication
Access Criteria: The request must be sent to the email address provided in the registration

REFERENCES:
- [Derived] Luchesi GLS, da Silva AKF, Amaral OHB, de Paula VCG, Jassi FJ. Effects of osteopathic manipulative treatment associated with pain education and clinical hypnosis in individuals with chronic low back pain: study protocol for a randomized sham-controlled clinical trial. Trials. 2022 Dec 30;23(1):1066. doi: 10.1186/s13063-022-07040-y. PMID 36581902